CLINICAL TRIAL: NCT02181699
Title: Phase 1 Study of KHK2823 in Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome.
Brief Title: Study of KHK2823 in Patients With Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Failed treatment response
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2823-001; 2013-003657-21 (EudraCT Number)
Record Dates: First submitted 2014-06-12; First posted 2014-07-04 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KHK2823 (Experimental): single agent KHK2823 administered at selected dose levels
  Interventions: Drug: KHK2823

INTERVENTIONS:
Drug: KHK2823 — single agent KHK2823

SUMMARY:
This is a first in human, non-randomized, open-label, dose escalation study to investigate the safety, pharmacokinetics, immunogenicity and pharmacodynamics of repeat doses of KHK2823.

DETAILED DESCRIPTION:
This is a Phase 1, multi-center, open-label, dose-escalation study of KHK2823 in adult patients with previously untreated AML who are not candidates for intensive remission induction therapy; relapsed/refractory AML for whom no other standard therapy is available or appropriate; or relapsed/refractory MDS who have received prior therapy with a hypomethylating agent, such as decitabine and azacitidine or who are not candidates to receive a hypomethylating agent, this would include high risk or transfusion-dependent low risk patients. Patients must have documented primary or secondary AML or MDS according to World Health Organization (WHO) criteria. Following the provision of signed informed consent, patients will be screened for entry into the study. The study consists of 2 parts. In Part 1, 3 to 6 patients per cohort will be enrolled sequentially in up to 7 dose-escalation cohorts to establish the MTD. KHK2823 will be administered once weekly. In Part 2, up to an additional 18 patients may be enrolled to further evaluate the safety, PK, PD, potential anti-leukemic activity of KHK2823.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years old with previously untreated AML who are not candidates for intensive remission induction therapy; relapsed/refractory AML for whom no other standard therapy is available or appropriate; or relapsed/refractory MDS who have received prior therapy with a hypomethylating agent or who are not candidates to receive a hypomethylating agent
* Histopathologically/cytologically documented primary or secondary AML, as defined by WHO criteria, or MDS, confirmed by pathology review at treating institution
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
* Life expectancy of at least 3 months

Exclusion Criteria:

* Histological diagnosis of acute promyelocytic leukemia (FAB Type M3)
* Clinically significant central nervous system leukemia
* Treatment of the underlying hematologic condition with systemic therapy during the treatment period, including any chemotherapy, radiation or investigational therapy, within 2 weeks prior to KHK2823 administration; or immunotherapy within 30 days prior to KHK2823 administration; with the exception of hydroxyurea (Hydrea®) for treatment of hyperleukocytosis, which must be discontinued at least 24 hours prior to the first dose of KHK2823

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability. | Assessed weekly for duration of treatment (anticipated minimum 8 weeks), plus 42 day follow up period

SECONDARY OUTCOMES:
Pharmacokinetics: Peak serum concentration (Cmax) Time to reach Cmax (tmax) Minimum serum concentration (Ctrough) Area under curve (AUC) Half-life (t1/2) Clearance (CL) Volume of distribution (Vd) Accumulation ratio (R) | Assessed during first 24 weeks of treatment, plus 42 day follow up period
Disease Response: overall response rate (ORR), overall survival (OS), event-free survival (EFS), relapse-free survival (RFS), progression-free survival (PFS) and disease-free survival (DFS) | Assessed every 8 weeks for duration of treatment (anticipated minimum 8 weeks), plus 14 day follow up period
Immunogenicity: anti-KHK2823 antibody | Assessed every 4 weeks for first 24 weeks of treatment, plus 42 day follow up period
  Measure of human anti-drug antibody
Pharmacodynamics: CD123+ | Assessed during first 24 weeks of treatment, plus 42 day follow up period
  Measure of KHK2823 target expression

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - University of Sussex, Royal Sussex County Hospital, Brighton
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's Institute of Oncology, Leeds
  - NIHR/Wellcome UCLH Clinical Research Facility University College Hospital London, London
  - St Bartholomew's Hospital, London
  - Northern Centre for Cancer Care, Freeman Road Hospital, Newcastle upon Tyne
  - Southampton General Hospital, Southampton